CLINICAL TRIAL: NCT00163904
Title: Can a Modified Fat Diet With Low Glycaemic Load Improve Insulin Sensitivity and Inflammatory Mediators in Overweight People With Chronic Heart Failure?
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12/05; Small Project Grant - T10513; Allied Health Grant - A10501
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2005-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Inflammatory mediators; insulin sensitivity; overweight; high monounsaturated diet
MeSH Terms: conditions — Heart Failure; Insulin Resistance; Overweight

INTERVENTIONS:
Behavioral: High mono-unsaturated fat/low carbohydrate diet
Behavioral: High carbohydrate/low fat diet

SUMMARY:
This study is looking at overweight patients with chronic heart failure (CHF), to compare the effects of a modified fat diet with a reduced glycaemic load (diet 1); and a conventional low fat, high carbohydrate diet (diet 2) on:

* insulin sensitivity (using the homeostasis model assessment [HOMA] model)
* lipid profile
* symptomatic status (6 minute walk distance and Heart Failure Quality of Life [HF QOL] Questionnaire)
* body weight
* inflammatory mediators (tumor necrosis factor [TNF] alpha, C-reactive protein [CRP], interleukin-6 [IL-6])

The hypotheses of this study are:

* Diet 1 will be associated with lower insulin resistance than diet 2.
* The lipid profile will be better in CHF patients on diet 1 than on diet 2.
* Patients on diet 1 will have a better symptomatic status than patients on diet 2.
* Diet 1 will maintain body weight in patients with CHF as well as diet 2.
* Diet 1 will suppress the expression of TNF-alpha, CRP and IL-6 more than diet 2.

DETAILED DESCRIPTION:
There is an increasing prevalence of chronic heart failure (CHF) in Western societies. In the last decade, progress has been made in understanding the neurohormonal involvement in the progression of the disease and consequently, new treatments have been developed although the mortality rate still remains high. Chronic heart failure is associated with marked insulin resistance as well as increasing plasma levels of pro-inflammatory markers such as Tumor Necrosis Factor-alpha (TNF-alpha) and Interleukin-6 (IL-6) with increasing severity of the disease. This has recently become an area of increased research interest. In CHF, insulin resistance may be present even when blood glucose levels appear normal. Independently of its influence on risk of arteriosclerosis, insulin resistance supports further progression of heart failure. Hyperinsulinaemia has also been found to worsen symptomatic status in CHF patients.

The introduction of beta-blockers in the treatment of CHF may have a beneficial effect on insulin resistance. However, so far tested drugs seem to have little influence on production of pro-inflammatory markers in CHF patients. The use of beta-blockers in the clinical setting is also associated with weight gain. While weight gain is of benefit to patients with cachexia, a common problem in CHF, it is problematic in CHF patients who are already overweight, particularly since obesity is known to be implicated in the development of insulin resistance. Because of this, it would seem to be beneficial to prevent further weight gain in those patients with heart failure who are not cachexic. Weight loss in these patients, however should also be prevented since obese patients with CHF appear to have the better prognosis. As change in body weight has important implications for disease progression, choice of dietary treatment is of particular importance in CHF patients. Ideally in CHF patients, we should be maintaining body weight while still attempting to reduce other coronary risk factors such as insulin resistance and atherogenic dyslipidemia.

Traditionally, diet for people with insulin resistance and other features of the metabolic syndrome has been based on a low fat, high carbohydrate dietary prescription. This has been questioned recently with emerging clear endorsement of diets that are restricted in saturated fat (< 10% of total energy [%E]) but by allowing higher amounts of monounsaturated fat (MUFA), also reduce the diet carbohydrate content and thus the glycaemic load. Metabolic studies in people with diabetes have shown that modified fat (high MUFA) diets are more effective than a low fat high carbohydrate diet in improving insulin resistance although no similar studies are yet available for people with heart failure.

Studies in people with diabetes have also indicated that modified fat (high MUFA) diets are clearly more beneficial than low fat diets in the effects on triacylglycerols and HDL cholesterol and they also favorably influence blood pressure, coagulation, endothelial activation, inflammation, and thermogenic capacity. Modified fat (high MUFA) diets therefore reduce heart disease risk. Moreover, when the energy density is controlled through inclusion of plenty of fruit and vegetables, modified fat (high MUFA) diets do not promote obesity. One final benefit is better acceptance and compliance long term.

ELIGIBILITY:
Inclusion Criteria:

* English speaking heart failure patients (New York Heart Association [NYHA] Classes 1 - 3) attending the Alfred Hospital outpatient clinic will be enrolled.

Exclusion Criteria:

* Patients will be excluded if they are below the healthy weight range (BMI < 25 kg/m2) or if they are morbidly obese (BMI > 35 kg/m2).
* Patients with heart failure NYHA Class 4 will be excluded due to their increased risk of developing cachexia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-01

PRIMARY OUTCOMES:
Body mass index (BMI)
Blood lipids
Inflammatory mediators
HOMA

SECONDARY OUTCOMES:
Heart Failure Quality of Life Questionnaire
6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Fiona J Adams, BSc. Grad Dip Diet, Principal Investigator — Dietition on Staff, Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia